CLINICAL TRIAL: NCT02795988
Title: A Phase 1b/2 Open-Label Study With Randomization in Phase 2 of IMU-131 HER2/Neu Peptide Vaccine Plus Standard of Care Chemotherapy in Patients With HER2/Neu Overexpressing Metastatic or Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction
Brief Title: A Study of IMU-131(HER-Vaxx) and Chemotherapy Compared to Chemotherapy Only in Patients With HER2 Positive Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Imugene Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMU.ACS.001
Record Dates: First submitted 2016-06-01; First posted 2016-06-10 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Gastrointestinal Neoplasms; Adenocarcinoma
Keywords: Secondary
MeSH Terms: conditions — Gastrointestinal Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Cisplatin; Fluorouracil; Capecitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Partially blinded - blinded central review of progression.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1b (Experimental): 10, 30, 50μg IMU-131 plus Cisplatin and either Fluorouracil (5-FU) or Capecitabine
  Interventions: Biological: IMU-131; Drug: Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and capecitabine.
- Phase 2 - IMU 131 plus chemotherapy (Experimental): 50 μg IMU-131 plus Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and Capecitabine.
  Interventions: Biological: IMU-131; Drug: Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and capecitabine.
- Phase 2 - Chemotherapy only (Experimental): Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and Capecitabine.
  Interventions: Drug: Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and capecitabine.

INTERVENTIONS:
Biological: IMU-131 — IMU-131 vaccine is a P467-CRM197 peptide antigen in PBS buffer and Montanide ISA 51 Sterile adjuvant
  Other Names: HER-Vaxx
  Arms: Phase 1b; Phase 2 - IMU 131 plus chemotherapy
Drug: Cisplatin and either Fluorouracil (5-FU) or Capecitabine or Oxaliplatin and capecitabine. — Chemotherapy will consist of: cisplatin by intravenous administration at 80 mg/m2 on the first day of each cycle and either 5-FU, 4000 mg/m2 CIV (administered as 1000 mg/m2/day as continuous infusion for 96 hours on days 1 to 4 of each cycle) or capecitabine for 14 days at 2000 mg/m2/day, orally (administered as 1000 mg/m2 twice daily morning and evening for a total of 2000 mg/m2/day on days 1 to 14 of each cycle), or (in Phase 2 only) oxaliplatin, by intravenous administration at 130 mg/m2 on Day 1 of each cycle and capecitabine for 14 days at 2000 mg/m2/day, orally (administered as 1000 mg/m2 twice daily morning and evening for a total of 2000 mg/m2/day on days 1 to 14 of each cycle).
  Other Names: Standard of Care Chemotherapy

SUMMARY:
The Phase 1b study is an open-label, multicenter dose escalation study designed to assess the safety, tolerability, immunogenicity and recommended phase 2 dose (RP2D) of IMU-131. The RP2D will be evaluated in the dose expansion Phase 2 study. The Phase 2 study is a randomized, open label comparison of IMU-131 plus standard of care chemotherapy versus standard of care chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been informed of the investigational nature of this study and has given written informed consent in accordance with institutional, local, and national guidelines;
2. Age ≥ 20 years old;
3. Life expectancy of at least 12 weeks;
4. Phase 1b: No prior chemotherapy or radiotherapy for advanced gastric or GEJ cancer within 6 months prior to Day 0; Phase 2: No prior chemotherapy or radiotherapy for advanced gastric or GEJ cancer within 3 months prior to Day 0;
5. Metastatic gastric or GEJ adenocarcinoma, or locally advanced disease not amenable to surgical resection;
6. HER2/neu overexpression (3+ by immunohistochemistry (IHC) or if IHC 2+ confirmed by fluorescent in situ hybridization [FISH] or chromogenic in situ hybridization [CISH]). Patients with IHC 2+ expression without confirmation of overexpression by fluorescent in situ hybridization [FISH] or chromogenic in situ hybridization [CISH]) may be included in Phase 1b with agreement of Imugene Limited;
7. Phase 1b: ECOG performance status 0-1; Phase 2: ECOG performance status 0-2;
8. At least one measurable lesion as defined by RECIST 1.1 criteria. Patients with non-measurable lesions may be included in Phase1b with agreement of Imugene Limited;
9. Adequate left ventricular ejection function at baseline, defined as LVEF > 50% by echocardiogram or MUGA scan (Multi Gated Acquisition Scan);
10. Adequate hematologic function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL;
11. Adequate liver function evidenced by bilirubin ≤ 1.5 x laboratory upper limit of normal [ULN], and ALT and AST ≤ 3 x laboratory ULN if no liver involvement or ALT and AST ≤ 5 times laboratory ULN with liver involvement;
12. Adequate renal function (creatinine ≤ 1.5 x laboratory ULN);
13. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
14. Male and female patients of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 28 days after the last dose of assigned treatment (see section 4.3 for details). A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

Exclusion Criteria:

1. Previous treatment with trastuzumab or any other HER2/neu targeting antibody or agent;
2. Continuous systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 4 weeks prior to first dose of study treatment. Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalents are permitted in the absence of active auto-immune disease;
3. Prior organ transplant;
4. Phase 1b: Patient not considered a candidate for 5-FU, capecitabine, or cisplatin chemotherapy; Phase 2: Patient not considered a candidate for 5-FU, capecitabine, cisplatin or oxaliplatin chemotherapy;
5. History of documented congestive heart failure; angina pectoris requiring antianginal medication; evidence of transmural infarction on ECG; poorly controlled hypertension; clinically significant valvular heart disease; high risk uncontrolled arrhythmias; or New York Heart Association (NYHA) class II heart disease;
6. If on warfarin (Coumadin®) or other vitamin K antagonists;
7. Concurrent active malignancy except for adequately controlled limited basal cell carcinoma of the skin;
8. Peripheral neuropathy or hearing loss of NCI CTCAE Grade > 2;
9. History of uncontrolled seizures, central nervous disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent, participation in the study, or adversely affecting compliance to study drugs;
10. Active infection requiring IV antibiotics;
11. Positive for human immunodeficiency virus (HIV) (HIV 1/2 antibodies) or active hepatitis B (HBsAg reactive) or active hepatitis C (HCV ribonucleic acid [RNA] qualitative) infection;
12. Pregnant or lactating females;
13. Major surgery within 4 weeks prior to study entry. Minor surgery (excluding diagnostic biopsy) within 1 week prior to study entry;
14. Has received a live-virus vaccination within 4 weeks of first study vaccination. Seasonal flu vaccines that do not contain live virus are permitted;
15. Current or recent (within 4 weeks of first IMU-131 vaccination) treatment with another investigational drug or participation in another investigational study.
16. Phase 2: Patients with a known diphtheria toxoid hypersensitivity.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- India (10):
  - City Cancer Center, Vijayawada, Andhra Pradesh
  - North East Cancer Hospital and Research Institute, Guwahati, Assam
  - Shetty's Hospital, Bengaluru, Karnataka
  - Curie Manavata Cancer Centre, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Victoria Hospital, Bangalore
  - MNJ Institute of Oncology and Regional Cancer Centre, Hyderabad
  - Tata Medical Centre, Kolkata
  - HCG NCHRI Cancer Centre, Nagpur
  - Regional Cancer Centre Indira Gandhi Institute of Medical Sciences, Patna
- ARENSIA Exploratory Medicine IMSP Institutul Oncologic, Chisinau, Moldova
- Serbia (4):
  - Oncology Institute of Vojvodina, Kamenitz, Južnobanatski Okrug
  - Institute for Oncology and Radiology of Serbia - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
- Taiwan (2):
  - National Cheng-Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
- Thailand (3):
  - Division of Medical Oncology, Department of Medicine, Prince of Songkla University, Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - National Cancer Institute of Thailand, Bangkok
  - Division of Oncology, Department of Internal Medicine, Faculty of Medicine, Chiang Mai University, Chiang Mai
- ARENSIA Exploratory Medicine LLC, Kapitanivka, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobias J, Maglakelidze M, Andric Z, Ryspayeva D, Bulat I, Nikolic I, Petrovic Z, Chawla T, Nagarkar R, Garner-Spitzer E, Zielinski CC, Chong LMO, Nixon B, Ede NJ, Yavrom S, Kundi M, Wiedermann U. Phase II Trial of HER-Vaxx, a B-cell Peptide-Based Vaccine, in HER2-Overexpressing Advanced Gastric Cancer Patients Under Platinum-Based Chemotherapy (HERIZON). Clin Cancer Res. 2024 Sep 13;30(18):4044-4054. doi: 10.1158/1078-0432.CCR-24-0742. PMID 39028916
- [Derived] Wiedermann U, Garner-Spitzer E, Chao Y, Maglakelidze M, Bulat I, Dechaphunkul A, Arpornwirat W, Charoentum C, Yen CJ, Yau TC, Tanasanvimon S, Maneechavakajorn J, Sookprasert A, Bai LY, Chou WC, Ungtrakul T, Drinic M, Tobias J, Zielinski CC, Chong L, Ede NJ, Marino MT, Good AJ. Clinical and Immunologic Responses to a B-Cell Epitope Vaccine in Patients with HER2/neu-Overexpressing Advanced Gastric Cancer-Results from Phase Ib Trial IMU.ACS.001. Clin Cancer Res. 2021 Jul 1;27(13):3649-3660. doi: 10.1158/1078-0432.CCR-20-3742. Epub 2021 Apr 20. PMID 33879458
- See also: Imugene (ASX: IMU) is a publicly-listed biotechnology company. — http://www.imugene.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 64 participants were enrolled in the study. Phase 1b, Phase 2, and Phase 2 extension parts enrolled separate participant populations.
Groups:
- Phase 1b: 10 μg IMU-131 Plus Chemotherapy: Participants received IMU-131 in intramuscular (IM) injections at a single dose level of 10 micrograms (μg) on Days 0, 14, 35, 98 and then every 12 weeks accompanied by chemotherapy every 21 days starting from Day 14. Chemotherapy included intravenous (IV) cisplatin and either Fluorouracil (5-FU) infusion or oral capecitabine.
- Phase 1b: 30 μg IMU-131 Plus Chemotherapy: Participants received IMU-131 in IM injections at a single dose level of 30 μg on Days 0, 14, 35, 98 and then every 12 weeks accompanied by chemotherapy every 21 days starting from Day 14. Chemotherapy included IV cisplatin and either 5-FU infusion or oral capecitabine.
- Phase 1b: 50 μg IMU-131 Plus Chemotherapy: Participants received IMU-131 in IM injections at a single dose level of 50 μg on Days 0, 14, 35, 98 and then every 12 weeks accompanied by chemotherapy every 21 days starting from Day 14. Chemotherapy included IV cisplatin and either 5-FU infusion or oral capecitabine.
- Phase 2: IMU-131 Plus Chemotherapy: Participants received IMU-131 in IM injections at dose level of 50 μg on Days 0, 14, 35, 77, and 140, then every 63 days until disease progression accompanied by chemotherapy every 21 days for up to 6 cycles starting from Day 14. Chemotherapy included one of the following treatments:
  * IV cisplatin and either 5-FU infusion or oral capecitabine.
  * IV oxaliplatin and oral capecitabine.
- Phase 2: Chemotherapy Only: Participants received chemotherapy every 21 days for up to 6 cycles starting from Day 14. Chemotherapy included one of the following treatments:
  * IV cisplatin and either 5-FU infusion or oral capecitabine.
  * IV oxaliplatin and oral capecitabine.
- Phase 2 Extension: IMU-131 100 μg: Participants received IMU-131 in IM injections at dose level of 100 μg on Days 0, 14, and 35, then every 63 days until disease progression accompanied by chemotherapy every 21 days for up to 6 cycles starting from Day 0. Chemotherapy included one of the following treatments:
  * IV cisplatin and either 5-FU infusion or oral capecitabine.
  * IV oxaliplatin and oral capecitabine.
- Phase 2 Extension: IMU-131 200 μg: Participants received IMU-131 in IM injections at dose level of 200 μg on Days 0, 14, and 35, then every 63 days until disease progression accompanied by chemotherapy every 21 days for up to 6 cycles starting from Day 0. Chemotherapy included one of the following treatments:
  * IV cisplatin and either 5-FU infusion or oral capecitabine.
  * IV oxaliplatin and oral capecitabine.
Period: Phase 1b
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Started | 3 | 6 | 5 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 6 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not Completed | 3 | 5 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 2 | 2 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Started | 0 | 0 | 0 | 19 | 17 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 18 | 14 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 19 | 17 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 17 | 17 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Phase 2 Extension
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Started | 0 | 0 | 0 | 0 | 0 | 7 | 7
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 7 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 7 | 7
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 5 | 6
Not completed — Other reasons | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population included all randomized participants.
Groups:
- Phase 1b: 10 μg IMU-131 Plus Chemotherapy: Participants received IMU-131 in IM injections at a single dose level of 10 μg on Days 0, 14, 35, 98 and then every 12 weeks accompanied by chemotherapy every 21 days starting from Day 14. Chemotherapy included IV cisplatin and either 5-FU infusion or oral capecitabine.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg | Total
Number analyzed (Participants) | 3 | 6 | 5 | 19 | 17 | 7 | 7 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Phase 1b, Phase 2, and Phase 2 Extension parts enrolled separate participant populations and are reported here separately.
  years
    Phase 1b: number analyzed (Participants) | 3 | 6 | 5 | 0 | 0 | 0 | 0 | 14
    Phase 1b | 51.0 (24.6) | 60.3 (9.8) | 57.4 (21.0) |  |  |  |  | 57.3 (16.7)
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 19 | 17 | 0 | 0 | 36
    Phase 2 |  |  |  | 64.4 (8.53) | 64.6 (10.31) |  |  | 64.5 (9.28)
    Phase 2 Extension: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 14
    Phase 2 Extension |  |  |  |  |  | 62.1 (15.19) | 69.7 (9.25) | 65.9 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Phase 1b, Phase 2, and Phase 2 Extension parts enrolled separate participant populations and are reported here separately.
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 6 | 5 | 0 | 0 | 0 | 0 | 14
    Phase 1b: Female | 2 | 2 | 1 |  |  |  |  | 5
    Phase 1b: Male | 1 | 4 | 4 |  |  |  |  | 9
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 19 | 17 | 0 | 0 | 36
    Phase 2: Female |  |  |  | 9 | 4 |  |  | 13
    Phase 2: Male |  |  |  | 10 | 13 |  |  | 23
    Phase 2 Extension: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 14
    Phase 2 Extension: Female |  |  |  |  |  | 1 | 2 | 3
    Phase 2 Extension: Male |  |  |  |  |  | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Phase 1b, Phase 2, and Phase 2 Extension parts enrolled separate participant populations and are reported here separately.
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 6 | 5 | 0 | 0 | 0 | 0 | 14
    Phase 1b: Hispanic or Latino | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: Not Hispanic or Latino | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: Unknown or Not Reported | 3 | 6 | 5 |  |  |  |  | 14
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 19 | 17 | 0 | 0 | 36
    Phase 2: Hispanic or Latino |  |  |  | 0 | 1 |  |  | 1
    Phase 2: Not Hispanic or Latino |  |  |  | 19 | 16 |  |  | 35
    Phase 2: Unknown or Not Reported |  |  |  | 0 | 0 |  |  | 0
    Phase 2 Extension: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 14
    Phase 2 Extension: Hispanic or Latino |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: Not Hispanic or Latino |  |  |  |  |  | 7 | 7 | 14
    Phase 2 Extension: Unknown or Not Reported |  |  |  |  |  | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Phase 1b, Phase 2, and Phase 2 Extension parts enrolled separate participant populations and are reported here separately.
  Participants
    Phase 1b: number analyzed (Participants) | 3 | 6 | 5 | 0 | 0 | 0 | 0 | 14
    Phase 1b: American Indian or Alaska Native | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: Asian | 3 | 4 | 2 |  |  |  |  | 9
    Phase 1b: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: Black or African American | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: White | 0 | 2 | 3 |  |  |  |  | 5
    Phase 1b: More than one race | 0 | 0 | 0 |  |  |  |  | 0
    Phase 1b: Unknown or Not Reported | 0 | 0 | 0 |  |  |  |  | 0
    Phase 2: number analyzed (Participants) | 0 | 0 | 0 | 19 | 17 | 0 | 0 | 36
    Phase 2: American Indian or Alaska Native |  |  |  | 0 | 0 |  |  | 0
    Phase 2: Asian |  |  |  | 3 | 0 |  |  | 3
    Phase 2: Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0 |  |  | 0
    Phase 2: Black or African American |  |  |  | 0 | 0 |  |  | 0
    Phase 2: White |  |  |  | 16 | 17 |  |  | 33
    Phase 2: More than one race |  |  |  | 0 | 0 |  |  | 0
    Phase 2: Unknown or Not Reported |  |  |  | 0 | 0 |  |  | 0
    Phase 2 Extension: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 14
    Phase 2 Extension: American Indian or Alaska Native |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: Asian |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: Native Hawaiian or Other Pacific Islander |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: Black or African American |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: White |  |  |  |  |  | 7 | 7 | 14
    Phase 2 Extension: More than one race |  |  |  |  |  | 0 | 0 | 0
    Phase 2 Extension: Unknown or Not Reported |  |  |  |  |  | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in the Reported AE section.
Time Frame: Up to approximately 7 months
Population: The Safety population included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy
Number analyzed (Participants) | 3 | 6 | 5
Participants | 3 | 6 | 5

2. Primary Outcome: Phase 2: Overall Survival (OS)
Description: OS was measured from date of randomization to date of death due to any cause.
Time Frame: Up to approximately 30 months
Population: The Intent-to-Treat population included all randomized participants.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only
Number analyzed (Participants) | 19 | 17
months | 13.90 [7.52 to 14.32] | 8.31 [6.01 to 9.59]
Statistical Analysis 1: Comparison: Phase 2: IMU-131 Plus Chemotherapy vs Phase 2: Chemotherapy Only; Test type: Superiority; p = 0.078, Log Rank — 1-sided p-value was calculated from Log-rank test stratified by factor tumor stage which used for randomization at screening; Cox proportional hazard regression model = 0.603, 80% CI 2-sided [0.380 to 0.957]

3. Primary Outcome: Phase 2 Extension: Number of Participants With AEs
Description: as for outcome 1
Time Frame: From date of first dose to date of last dose plus 30 days (Up to 24 months)
Population: The Safety population included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 7 | 7
Participants | 7 | 5

4. Secondary Outcome: Phase 2 and Phase 2 Extension: Progression-Free Survival (PFS)
Description: PFS was measured from randomization to date of earliest progressive disease (PD) based on blinded central review according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, or to date of death from any cause.
Time Frame: Up to approximately 30 months
Population: The ITT Population included all randomized participants.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 19 | 17 | 7 | 7
months | 6.93 [5.59 to 9.86] | 6.01 [2.17 to 8.31] | 5.03 [1.38 to 9.89] | 8.34 [5.52 to 8.34]

5. Secondary Outcome: Phase 2 and Phase 2 Extension: Time to Progression (TTP)
Description: TTP was measured from randomization to date of earliest PD based on blinded central review according to RECIST 1.1 criteria.
Time Frame: Up to approximately 30 months
Population: The ITT Population included all randomized participants.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 19 | 17 | 7 | 7
months | 6.93 [5.59 to 9.86] | 8.44 [8.44 to NA] — Upper Confidence Interval (CI) not reached due to insufficient number of events | 5 [4.1 to 8.9] | 5.5 [3.5 to 7.5]

6. Secondary Outcome: Phase 2 and Phase 2 Extension: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR), or stable disease according to RECIST 1.1 after randomization/enrollment date.
Time Frame: Up to approximately 30 months
Population: The Full Analysis Set (FAS) included all randomized participants who received any amount of study treatment.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 18 | 14 | 7 | 7
percentage of participants | 77.8 [63.20 to 87.70] | 71.4 [54.40 to 84.00] | 71.4 [47.20 to 87.50] | 85.7 [62.20 to 95.60]

7. Secondary Outcome: Phase 2 and Phase 2 Extension: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants with a BOR of CR or PR according RECIST 1.1 after randomization/enrollment date.
Time Frame: Up to approximately 30 months
Population: The FAS included all randomized participants who received any amount of study treatment. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 18 | 14 | 7 | 7
percentage of participants | 38.9 [25.70 to 53.90] | 50.0 [33.80 to 66.20] | 42.9 [22.60 to 65.80] | 71.4 [47.20 to 87.50]

8. Secondary Outcome: Phase 2 and Phase 2 Extension: Duration of Response (DOR)
Description: DOR was defined as the time from the earliest date when a tumor response of CR or PR was observed until the date of first occurrence of disease progression which assessed by the blinded central reviewer or death (due to any reason).
Time Frame: Up to approximately 30 months
Population: All randomized participants with a BOR of CR or PR
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 7 | 7 | 3 | 5
months | 7.10 [2.79 to NA] — Upper 80% CI not reached due to insufficient number of events | 4.40 [4.07 to NA] — Upper 80% CI not reached due to insufficient number of events | 3.65 [2.92 to NA] — Upper 80% CI not reached due to insufficient number of events | 5.59 [1.12 to 5.59]

9. Secondary Outcome: Phase 2 and Phase 2 Extension: Percentage Change From Baseline in Tumor Size
Description: Change in tumor size (CTS) was measured as the sum of diameters based on blinded central review according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1).
Time Frame: Baseline up to approximately 30 months
Population: The ITT Population included all randomized participants. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure.
Measure: Median (80% Confidence Interval); unit: percentage change from baseline
Arm/Group | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 15 | 13 | 7 | 6
percentage change from baseline | -22.4 [-39.4 to -19.7] | -34.4 [-34.6 to -16.9] | -43.1 [-53.7 to -38.0] | -36.8 [-47.7 to -32.2]

10. Secondary Outcome: Phase 2 Extension: OS
Description: OS was measured from date of randomization to date of death due to any cause.
Time Frame: Up to 24 months
Population: The FAS included all randomized participants who received any amount of study treatment.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
Number analyzed (Participants) | 7 | 7
months | 18.27 [5.03 to 19.84] | 9.36 [4.40 to NA] — Upper 80% CI not reached due to insufficient number of events

ADVERSE EVENTS:
Time Frame: Up to approximately 30 months
Arm/Group | Phase 1b: 10 μg IMU-131 Plus Chemotherapy | Phase 1b: 30 μg IMU-131 Plus Chemotherapy | Phase 1b: 50 μg IMU-131 Plus Chemotherapy | Phase 2: IMU-131 Plus Chemotherapy | Phase 2: Chemotherapy Only | Phase 2 Extension: IMU-131 100 μg | Phase 2 Extension: IMU-131 200 μg
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/6 | 1/5 | 17/19 | 17/17 | 5/7 | 6/7
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/6 | 3/5 | 2/19 | 5/17 | 0/7 | 2/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 18/19 | 15/17 | 7/7 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: 10 μg IMU-131 Plus Chemotherapy (N=3) | Phase 1b: 30 μg IMU-131 Plus Chemotherapy (N=6) | Phase 1b: 50 μg IMU-131 Plus Chemotherapy (N=5) | Phase 2: IMU-131 Plus Chemotherapy (N=19) | Phase 2: Chemotherapy Only (N=17) | Phase 2 Extension: IMU-131 100 μg (N=7) | Phase 2 Extension: IMU-131 200 μg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: 10 μg IMU-131 Plus Chemotherapy (N=3) | Phase 1b: 30 μg IMU-131 Plus Chemotherapy (N=6) | Phase 1b: 50 μg IMU-131 Plus Chemotherapy (N=5) | Phase 2: IMU-131 Plus Chemotherapy (N=19) | Phase 2: Chemotherapy Only (N=17) | Phase 2 Extension: IMU-131 100 μg (N=7) | Phase 2 Extension: IMU-131 200 μg (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 0 | 3 | 5 | 2 | 0
Anaemia folate deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2 | 5 | 3 | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 3 | 4 | 1 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 3 | 2 | 2
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 3 | 1 | 5 | 2 | 1 | 3
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 1 | 1 | 1 | 1 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Administration site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 2 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 1 | 2 | 1 | 2 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1 | 4 | 2 | 0
Protein total increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 2 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 2 | 5 | 1 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT02795988/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT02795988/SAP_001.pdf